CLINICAL TRIAL: NCT03865654
Title: Individualizing Surveillance Mammography for Older Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rachel Freedman, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-001; 1R21CA227615-01A1 (NIH)
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Results first posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surveillance Mammography Communication Tool (Experimental): * Conduct 30 telephone-based patient interviews
  * 4-6 focus groups with oncologists and primary care providers (PCs) to learn their perceptions and thoughts about when to stop surveillance mammography
  * Perform cognitive testing of the communication tool
  Interventions: Other: Communication Tool

INTERVENTIONS:
Other: Communication Tool — Summarizes recommendations for clinicians and patients for surveillance mammography and follow-up care for breast cancer survivors

SUMMARY:
This research is being conducted to develop consensus on surveillance mammography and follow-up for breast cancer survivors who are age ≥75.

DETAILED DESCRIPTION:
The investigators will develop a communication tool that summarizes recommendations for clinicians and patients for surveillance mammography and follow-up care for breast cancer survivors age ≥75. Developing expert-panel recommendations, examining clinician and patient attitudes towards these recommendations, and testing a strategy for communication of expert recommendations on mammography cessation through direct engagement of specialists, primary care clinicians (PCs), and patients.

This is a multi-step study, the investigators will build on prior steps to develop consensus on surveillance mammography and follow-ups for breast cancer survivors who are age >= 75.

This study includes a physician focus group.

ELIGIBILITY:
Inclusion Criteria:

* Female gender, given that screening guidelines do not exist for men
* Receiving part or all of their care at DFCI
* Ages 75-79 (approximately 15 patients)
* Age ≥80 (approximately 15 patients)
* History of stage 0-II breast cancer

  -≥1 Charlson comorbidity present72, defined as one of the following:
  * Diabetes
  * Liver disease
  * History of or other active malignancy other than non-melanoma skin cancers
  * HIV or AIDS
  * Chronic kidney disease
  * History of myocardial infarction and/or congestive heart failure
  * Chronic lung disease (emphysema/chronic bronchitis/chronic obstructive pulmonary disease [COPD], interstitial lung disease)
  * Peripheral vascular disease
  * Cerebrovascular disease (history of TIA or stroke)
  * Dementia
  * Hemiplegia/paralysis
  * Connective tissue disorder
* Underwent breast conserving surgery for treatment of this cancer
* Completed all active breast cancer therapy >3 months prior to enrollment (i.e. any chemotherapy, trastuzumab, radiation). Ongoing hormonal therapy or enrollment in survivorship clinical trials (aspirin, exercise, etc) is allowed.
* English-speaking and reading (for this initial work)
* Aim 1.1. Cognitive testing of the communication tool. The criteria for this are intentionally more flexible than in other aims, as we are simply working to initially test the tool and its readability and understandability. Patients will be eligible to cognitively test the tool if they meet the following criteria:
* Female gender
* Previous diagnosis of breast cancer
* Age ≥75
* Receive some/all care at Dana-Farber Cancer Institute
* English speaking-reading
* Aim 1.2. Pilot testing the communication tool in clinic.
* Previous diagnosis of stage 0-II breast cancer
* Receive some/all care at Dana-Farber Cancer Institute (main campus or St. Elizabeth's site)
* Completed any active breast cancer therapy > 3 months prior to enrollment (i.e. any chemotherapy, trastuzumab, radiation). Ongoing hormonal therapy or enrollment in survivorship clinical trials (aspirin, exercise, etc) is allowed.
* Age ≥75
* Had breast-conserving surgery to treat this cancer

  -≥1 the following comorbid conditions72 present, defined as the following:
  * Diabetes
  * Liver disease
  * History of or other active malignancy other than non-melanoma skin cancers
  * HIV or AIDS
  * Chronic kidney disease
  * History of myocardial infarction and/or congestive heart failure
  * Chronic lung disease (COPD, interstitial lung disease)
  * Peripheral vascular disease
  * Cerebrovascular disease (history of TIA or stroke)
  * Dementia
  * Hemiplegia/paralysis
  * Connective tissue disorder
* Provider does not opt out of the patient's enrollment via email notification
* Blessed Orientation Memory Concentration (COMC) score is <10 and capacity is met73 (see Appendix A for BOMC scale)
* Providers of participating patients will be sent a one-time survey but there are no other eligibility for providers to participate in this other than their patient participated
* English speaking and reading

Exclusion Criteria:

* Are unable to consent
* Who do not read and write English (for this initial pilot)

Min Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Freedman, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Freedman RA, Revette AC, Gagnon H, Perilla-Glen A, Kokoski M, Hussein SO, Leone E, Hixon N, Lovato R, Loeser W, Lin NU, Minami CA, Canin B, LeStage B, Faggen M, Poorvu PD, McKenna J, Ruddy KJ, Keating NL, Schonberg MA. Acceptability of a companion patient guide to support expert consensus guidelines on surveillance mammography in older breast cancer survivors. Breast Cancer Res Treat. 2022 Sep;195(2):141-152. doi: 10.1007/s10549-022-06676-3. Epub 2022 Jul 30. PMID 35908120

RESULTS

PARTICIPANT FLOW:
Groups:
- Surveillance Mammography Communication Tool: * Conduct 30 telephone-based patient interviews
  * 4-6 focus groups with oncologists and primary care providers (PCs) to learn their perceptions and thoughts about when to stop surveillance mammography
  * Perform cognitive testing of the communication tool
  Communication Tool: Summarizes recommendations for clinicians and patients for surveillance mammography and follow-up care for breast cancer survivors
Period: Overall Study
Arm/Group | Surveillance Mammography Communication Tool
Started | 45
Completed | 40
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Surveillance Mammography Communication Tool
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Intentions for Mammography in the Next Year
Description: Survey measure on whether mammography will be done or not
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Surveillance Mammography Communication Tool
Number analyzed (Participants) | 40
Participants
  Intention to undergo mammogram | 39
  Intention to not undergo mammogram | 1

2. Secondary Outcome: Rate of Satisfaction
Description: Survey asking about satisfaction with the tool
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Surveillance Mammography Communication Tool
Number analyzed (Participants) | 40
Participants
  Tool was very, somewhat, or a little helpful | 31
  Tool was not help | 6
  Did not respond | 3

3. Secondary Outcome: Preferred Decision-making Role
Description: Survey on preferred decision-making style
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Surveillance Mammography Communication Tool
Number analyzed (Participants) | 45
Participants
  I prefer to make the final decision. | 14
  I prefer to make the final decision after seriously considering my health care provider's opinion. | 15
  I prefer that my health care provider and I share responsibility for deciding . | 13
  I prefer that my health care provider makes the final decision, but seriously considers my opinion. | 3

ADVERSE EVENTS:
Time Frame: Not applicable- no adverse events for this survey-based study
Description: Not applicable, no adverse events for this survey-based study
Arm/Group | Surveillance Mammography Communication Tool
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT03865654/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT03865654/SAP_001.pdf